CLINICAL TRIAL: NCT01737060
Title: Clinical Investigation for Fractures of the Proximal Humerus in Elderly Patients. A Randomized Study of Two Surgical Treatments: Reverse Total Shoulder Arthroplasty Versus Angular Stable Device Philos
Brief Title: Displaced Proximal Humeral Fractures: Delta Prothesis or Philos Plate?
Acronym: DELPHI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Sykehuset Telemark (Other Government); Sykehuset Asker og Baerum (Other); Sykehuset Ostfold (Other); Helse Forde (Other); Sykehuset i Vestfold HF (Other); Diakonhjemmet Hospital (Other)
Responsible Party: Principal Investigator, Tore Fjalestad, MD PhD Senior Consultant, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RTSA s422
Record Dates: First submitted 2012-11-20; First posted 2012-11-29 (Estimated); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Proximal Humeral Fractures, AO/OTA (2007) Group B2 and C2
Keywords: Reversed prosthesis, Philos, Severe displaced
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Angular stable plate Philos (Active Comparator): Open Reduction and Osteofixation with Philos plate and TiCron cerclages
  Interventions: Device: Reverse total shoulder arthroplasty
- Reverse Total Shoulder Artroplasty (Experimental): Intervention group
  Interventions: Device: Reverse total shoulder arthroplasty

INTERVENTIONS:
Device: Reverse total shoulder arthroplasty
  Other Names: Delta Xtend shoulder proshesis

SUMMARY:
To investigate the assumption that reversed shoulder prosthetic replacement will give a better functional outcome compared to open reduction and internal fixation with an angular stable plate in displaced proximal humeral fractures. Short name: The DelPhi trial.

DETAILED DESCRIPTION:
Reversed total shoulder artroplasty (RTSA) equals Delta Xtend reversed total shoulder prosthesis.

Angular stable plate means Proximal humerus plate (Philos)

ELIGIBILITY:
Inclusion Criteria:

Patient admitted in hospital with a displaced three- or four part proximal humerus fracture of OTA / AO group 11-B2 or 11-C2 (displaced fracture of extra-articular or articular, bifocal type). The subgroups -.1, -.2 and -.3 will be included for both B2 and C2 groups, provided severe displacement: This is defined as a mal-position of at least 45º of angular deviation in valgus or 30º in varus in true frontal projection, regardless of whether the fracture is impacted or not, or less than 50% contact between humeral head and the metaphyseal part of the shaft. The greater or lesser tubercle displaced at least 10 mm.

Exclusion Criteria:

Patient younger than 65 years or older than 85 years, previous history of injury or illness of the injured shoulder, injuries of other parts of the humerus or the contra-lateral upper extremity, alcohol- or drug abuse, dementia, neurological diseases, or severe cardiovascular or lung diseases that would contraindicate surgery. Patients have to understand the Norwegian language and be compliant to rehabilitation and follow-ups.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 124 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Constant Shoulder Score | 5 years
  Follow-up will be at 3-6-12 months and 2-5 years.

SECONDARY OUTCOMES:
Oxford Shoulder score | 5 years
  Follow-up will be at 3-6-12 months and 2-5 years.

OTHER OUTCOMES:
15D Quality of Life score | 5 years
  Follow-up will be at 3-6-12 months and 2-5 years.
Health Economics | 5 years
  Follow-up will be at 3-6-12 months and 2-5 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Result] Fjalestad T, Iversen P, Hole MO, Smedsrud M, Madsen JE. Clinical investigation for displaced proximal humeral fractures in the elderly: a randomized study of two surgical treatments: reverse total prosthetic replacement versus angular stable plate Philos (The DELPHI-trial). BMC Musculoskelet Disord. 2014 Sep 28;15:323. doi: 10.1186/1471-2474-15-323. PMID 25261913
- [Result] Fraser AN, Bjordal J, Wagle TM, Karlberg AC, Lien OA, Eilertsen L, Mader K, Apold H, Larsen LB, Madsen JE, Fjalestad T. Reverse Shoulder Arthroplasty Is Superior to Plate Fixation at 2 Years for Displaced Proximal Humeral Fractures in the Elderly: A Multicenter Randomized Controlled Trial. J Bone Joint Surg Am. 2020 Mar 18;102(6):477-485. doi: 10.2106/JBJS.19.01071. PMID 31977825
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196
- [Derived] Bones I, Karlberg AC, Liljeholm M, Fraser AN, Madsen JE, Fjalestad T. Pegs not superior to screws for fixation of fractures of the proximal humerus. J Orthop Surg Res. 2022 Feb 2;17(1):66. doi: 10.1186/s13018-022-02947-3. PMID 35109905
- See also: Trial website for patients, their relatives and health workers — https://oslo-universitetssykehus.no/avdelinger/ortopedisk-klinikk/ortopedisk-avdeling-ulleval/seksjon-for-ortopedisk-traumatologi-ulleval/brudd-i-ovre-del-av-overarmsbeinet-proksimale-humerus-delphistudien